CLINICAL TRIAL: NCT01001156
Title: Effects of the Breathing Muscular Training to Volume and the Pressure in MIP and MEP of Institutionalized Elderly
Brief Title: Effects of the Breathing Muscular Training of Institutionalized Elderly
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Universidade Camilo Castelo Branco (Other)
Responsible Party: Marilia de Andrade Fonseca, Castelo Branco University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 0043-2008
Record Dates: First submitted 2009-10-21; First posted 2009-10-23 (Estimated); Last update posted 2009-10-23 (Estimated); Status verified 2009-10

CONDITIONS: In Brazil, Which Has an Increasing Number of Elderly People.; The Physiological Alterations of Aging Are Systemic.
Keywords: Aged; Breathing Muscles; Strength Muscles; Institution of long Permanence for elderly
MeSH Terms: interventions — Aging

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Other: Comparison of different breathing muscular training — Three times per week for ten weeks, thirty minutes.
  Other Names: Aged, Breathing Muscles, Strength Muscles.

SUMMARY:
The purpose of this study was to use associated breathing exercises the incentive inspiratory of load lineal pressoric, Threshold® IMT, or of load pressoric alinear, Voldyne®, in institutionalized elderly, comparing the effect of the same ones in the training of the breathing musculature, for the increment of the muscular strength, expressed by the maximum breathing pressures (MIP and MEP).

From the total number of admitted people (n = 52), 12 individuals were excluded: one by appearance of cognitive deficit, one by death (stroke), one by visual deficit (glaucoma) and twelve by failure to continue the training. After selecting the sample, the 37 participants were randomly divided into three different groups: the Threshold Group (TG; n = 13, age = 70. 93 ± 8.41 years old, BMI = 24.06 ± 3.69 kg/m²), the Voldyne Group (VG; n = 12, age = 70.54 ± 7. 73 years-old, BMI = 27.17 ± 5.66 kg/m²) and the Control Group (CG; n= 12, age = 73. 92 ± 7.28 years-old, BMI = 24.80 ± 5.42 kg/m²). The TG and VG received treatment with respiratory exercises and Threshold and Voldyne muscular training, respectively. The CG received only respiratory exercises.

DETAILED DESCRIPTION:
The physiologic alterations of the aging are systemic and they seem to be more evident in the institutionalized elderly. The advanced age is associated to the decrease of the force of the skeletal muscles, as well as the one of the muscles respiratory. In the breathing system happen important muscle-skeletal alterations, interfering in the mechanics ventilatory. The changes in the compliance of the thoracic wall and of the lung stcruture resulting in imprisonment of air, air-trapping ", increasing the breathing work simultaneously the and functional residual capacity (FRC) with consequent decrease of the pressure maximum expiratory. Also the decreases of the pick of flow expiratory and changes in the curve flow-volume contributing to the closing of the outlying aerial roads. This way the breathing muscular function will be strongly harmed and correlated with the state nutritional and it forces muscular outlying. Besides, modifications in the curvature of the diaphragm, with a negative effect for the capacity to generate muscular force, collaborating for the decrease inspiratory.

The participant was completely evaluated, including personal information, medical history and a physical examination.

Measurement of Translation provided gratis.

MIP and MEP: Before and after the respiratory muscle training, inspiratory and expiratory strength were evaluated and analysed through the maximum inspiratory pressure (MIP) and maximum expiratory pressure (MEP), respectively. This was measured using a device called a vacuum manometer (analogical with operational intervals of -120 to + 120 cmH2O, Critical Med/USA-2002 and display with scale intervals of 4 cmH2O). During MIP measurements, a nasal clip was used, which prevented air from escaping during the evaluation. In MIP measurements, the mouth and oropharynx can create negative pressure that can alter the results depending on whether the glottis opens (correct form) or closes (improper form). To prevent this interference of the orofacial musculature in the MIP measurements, an escape orifice was placed in the measurement instrument. This orifice relieved the pressure without significantly affecting the pressure produced by the respiratory muscles. Five tests were carried out to get three acceptable measures (i.e., duration of at least 2 seconds and an absence of emptying).

Acceptable tests were required to have at least two reproducible measurements (a maximum difference of 5% between the two maxima). A rest of at least one minute between tests was used for better equalization of the volumes and (consequently) the attainment of maximum pressures. To measure MEP, the patient was instructed to inhale until reaching total pulmonary capacity (TPC) and to carry through a supported expiratory effort down to the residual volume (RV). A seated position was used when measuring both MIP and MEP.

Threshold Group Training: after the measurement of the initial MIP and MEP (pre-training), the elderly individuals of the TG were submitted to a respiratory exercise program. The research of Ide et al. (2007) showed that this program contributes to an increase in chest expansion in healthy elderly people. The program was composed of the following exercises: active/resistance exercise of horizontal adduction-abduction and flexion-extension of the shoulder joint; active/resistance exercise of anterior flexion associated with rotation of the trunk and lateral flexion of the trunk; active/resistance exercise of lateral rotation of the trunk; active/resistance exercise to put the superior members above the head. The relaxation protocol consisted of inspiration and deep expiration without the accompaniment of other movements. After training, the Threshold® IMT (Respironics USA - 2004) was used. This device is commercially offered in the form of a transparent plastic cylinder; at one end is a valve that is kept closed for the positive pressure by a spring, while at the other end is a nipple. The valve blocks the aerial flow until the patient generates inspiratory pressure sufficient to overcome the spring.

The utilization of Threshold in this research began with a gradual load, starting with 50% of the MIP of each individual and increasing 10% per week until the fourth week. From the fifth week on, this was increased by 5% until 100% was reached in the eighth week or the maximum pressure value of the Threshold IMT (41 cmH2O) was reached. Thereafter, this value was kept constant in the final two weeks. The sessions lasted 20 minutes and consisted of seven series of strengthening (2 minutes each) with an interval of 1 minute between the series; sessions were conducted three times per week for ten weeks.

In the use of this training program, all the elderly individuals had been evaluated separately and trained in a group with individualized attention.

Voldyne Group Training: The same respiratory exercises used in the TG were used in the VG.

The maximum inspiratory sustentation technique (MIS) using the Voldyne mobilizes great pulmonary volumes and thereby increases the intra-alveolar pressure until the end of the supported inspiration. The increase in the intra-alveolar pressure is directly proportional to the contractile strength of the respiratory muscles (diaphragm and accessories), thus justifying the fact that intense muscular activity is required to reach the total pulmonary capacity (TPC) and to support inspiration at this level.

The use of EI (Voldyne®) incentive spirometry as muscular training in elderly people and as a basis for physiotherapy followed some guidelines. The patient's trunk was positioned at 30º relative to the horizontal plane, providing more diaphragmatic conscription. The device was positioned vertically. The volume indicator was visible to the patient to provide visual biofeedback. The patient was instructed to carry out a slow and deep inspiration until reaching TPC from the functional residual capacity (FRC). Slow inspiration favours a laminar flow. A sustentation of the maximum inspiration of around three seconds was recommended. Expiration occurred normally until the FRC was reached. During the use of Voldyne, patient hyperventilation was avoided. Intervals of 60 seconds between the inspiration support maxima were recommended 11. The elderly subjects received a verbal command to initiate a new inspiration. In this study, the Voldyne was used for 20 minutes, that is, 40 repetitions with 2 repetitions per minute. The procedure lasted 10 weeks at a frequency of three times per week. The group was supervised intermittently during the twenty minutes to ensure that hyperventilation was not occurring.

Control Group Training: This group received only respiratory exercises. The exercises was composed of the following exercises: active/resistance exercise of horizontal adduction-abduction and flexion-extension of the shoulder joint; active/resistance exercise of anterior flexion associated with rotation of the trunk and lateral flexion of the trunk; active/resistance exercise of lateral rotation of the trunk; active/resistance exercise to put the superior members above the head. The relaxation protocol consisted of inspiration and deep expiration without the accompaniment of other movements.

Statistical Treatment:The average and standard deviation (av ± sd) were calculated for age, body mass index, maximum respiratory pressure and functional autonomy. The normality of the sample was evaluated by the Shapiro-Wilk test and the homogeneity of the variance by the test of Levene. For the within-groups analysis variables, the parametric Student's t test or Wilcoxon was used when appropriate (for homogeneous or heterogeneous distribution of the data, respectively). For the between-groups evaluation, the nonparametric Kruskal-Wallis test was used followed by the Mann-Whitney multiple comparisons test. The statistical significance level adopted was p < 0.05. Excel and the SPSS v14.0 statistical package program were used to evaluate the data.

ELIGIBILITY:
Inclusion Criteria:

* The elderly individuals were required to be in good physical and cognitive condition to be considered for the study

Exclusion Criteria:

* Eliminated participation by those who had acute-phase infections of the cardio-respiratory system and those who did not have a satisfactory cognitive level to understand the evaluation tests and the exercises performed in the treatment programs.
* Also excluded were people who presented skeletal muscle and neurological sequel, presented metabolic syndromes or failed to adhere to the training program for more than one week.

Ages: 60 Years to 82 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2008-10; Primary Completion 2008-12 (Actual); Study Completion 2009-05 (Actual)

PRIMARY OUTCOMES:
Maximum inspiratory pressure (MIP) and maximum expiratory pressure (MEP) in cmH2O | One minute

SECONDARY OUTCOMES:
Before and after the respiratory muscle training, inspiratory and expiratory strength were evaluated and analysed through the maximum inspiratory pressure (MIP) and maximum expiratory pressure (MEP), respectively. | Ten weeks

CONTACTS AND LOCATIONS:
Overall Officials: Marilia A. Fonseca, Esp., Principal Investigator — Universidaade Castelo Branco; Samaria A. Cader, Dr., Study Director — Laboratory of Human Kinetics Bioscience from Castelo Branco University - LABIMH-UCB/Rio de Janeiro - RJ- Brazil; Silvia C. Bacelar, Dr., Study Chair — National Institute of Cancer (INCA) - Rio de Janeiro - RJ - Brazil; Elirez B. Silva, Dr., Study Chair — Gama Filho University (UGF) - Rio de Janeiro - RJ - Brazil; Silvânia O. Leal, Esp., Study Chair — Laboratory of Human Kinetics Bioscience from Castelo Branco University - LABIMH-UCB/Rio de Janeiro - RJ- Brazil; Estelio M. Dantas, Phd., Study Director — Laboratory of Human Kinetics Bioscience from Castelo Branco University LABIMH-UCB/ Rio de Janeiro- RJ- Brazil
Locations (1):
- Marilia de Andrade Fonseca, Rio de Janeiro, Rio de Janeiro, Brazil

REFERENCES:
- [Result] Hill K, Jenkins SC, Philippe DL, Cecins N, Shepherd KL, Green DJ, Hillman DR, Eastwood PR. High-intensity inspiratory muscle training in COPD. Eur Respir J. 2006 Jun;27(6):1119-28. doi: 10.1183/09031936.06.00105205. PMID 16772388
- See also: Comparative study of elderly inpatients clinically diagnosed with community-acquired pneumonia, with or without radiological confirmation. — http://www.scielo.br/scielo.php?script=sci_arttext&pid=S1806-37132007000300007&lng=pt.doi:10.1590/S1806-37132007000300007